CLINICAL TRIAL: NCT02380599
Title: A Comparative Study of the Effects of Mid-Thoracic Spinal Manipulation and Spinal Mobilization on Heart Rate Variability
Brief Title: A Study of the Effects of Mid-Thoracic Spinal Manipulation and Spinal Mobilization on Heart Rate Variability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mount St. Mary's College, Los Angeles, CA (Other)
Responsible Party: Principal Investigator, Derrick Sueki, Principal Investigator, Mount St. Mary's College, Los Angeles, CA
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: MountSMCLA 3
Record Dates: First submitted 2015-02-28; First posted 2015-03-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Physiology of Manipulation / Mobilization in Healthy Adults
Keywords: Spinal Manipulation; Mobilization; Autonomic Nervous System
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Group (Experimental): Crossover assignment of mid-thoracic spinal manipulation, spinal mobilization, or sham ultrasound
  Interventions: Other: Spinal Manipulation; Other: Spinal Mobilization; Other: Sham Ultrasound

INTERVENTIONS:
Other: Spinal Manipulation — Mid-thoracic spinal manipulation to T3-5 region
Other: Spinal Mobilization — Mid-thoracic spinal mobilization to T3-5 region
Other: Sham Ultrasound — Sham ultrasound to T3-5 region

SUMMARY:
Spinal mobilization and spinal manipulation are common techniques utilized in the field of physical therapy. Despite their common utility, little is known about the physiological mechanisms underlying the changes experienced following the interventions. Recent research suggests that neurological mechanisms may be involved in the post interventional changes, but research supporting this view is still evolving. Therefore, this study will explore whether there is a neurophysiological difference between spinal manipulation and spinal mobilization techniques. The neurophysiological difference will be measured by monitoring heart rate variability, a cardiovagal indicator of autonomic nervous system activity. The primary hypotheses of this study are three-fold, first that spinal manipulation will result in a change in heart rate variability that is different then sham intervention. Second, spinal mobilization will result in a change in heart rate variability that is different then sham intervention. Finally, the investigators hypothesize that spinal mobilization and spinal manipulation will produce different changes in heart rate variability.

DETAILED DESCRIPTION:
This study will utilize a crossover design to study autonomic nervous system responses in healthy subjects. Prior to commencing data collection, Institutional Review Board approval has been obtained from the Mount St. Mary's College Committee for the Protection of Human Subjects. Once obtained subjects will be recruited from faculty, students, and staff of the College. A snowball methodology will be used to recruit friends, family, and acquaintances of these initial connections. To be included in this study, candidates must be between the age of 18 and 55 years of age. They must not have pain in any area of their body that is chronic in nature (has been present for greater then three months). Subjects who are pregnant or have a history of spinal surgery will be excluded from participation in this study. All subjects who fulfill the inclusion and exclusion criteria will be informed of the intent, methods and risks associated with the study and given an opportunity to ask questions. Following this information session, and if agreeing to participate in the study, subjects will be asked to fill out the attached informed consent form. All subjects will be notified and given the opportunity to withdrawal from the study at any time without repercussions.

Once accepted into the study, subjects will fill out a personal history questionnaire to gather demographic information such as age, medical history, gender, and current pain levels. The subject will also be asked to fill out the General Anxiety Disorder 7-Item Scale Questionnaire. Once collected, subjects will be assigned a confidential subject number and all personal identifiers will be removed from subject information. All data will be scanned and stored in a personal computer that is password protect. Also at this time, subjects will be randomly assigned to a treatment group. Since this is a crossover design, all subjects will receive all interventions, but the order of these interventions will be predetermined and randomized.

At this point, subjects will be taken to a quiet room located within the Department of Physical Therapy. This room is used as a lab and data collection room and has a physical therapy treatment table. The subject will be asked to lie prone on the table and an electrocardiographic recording sensory will be placed upon each wrist (two total). This sensory will feed data regarding heart rate to a laptop computer that will be collected using the Biocomm HRV Live! Heart Rate Variability (HRV) Data Acquisition program. Once the strength and stability of the signal is verified, the subject will be instructed to rest quietly for five minutes in order to gather baseline heart rate data. Following this five-minute timeframe, the subject will receive one of three interventions based upon the previously mentioned randomization process. The three interventions utilized in the study will be a posterior to anterior spinal manipulation delivered to T4-5 spinal segment, posterior to anterior spinal mobilization applied to the T4-5 spinal segment for 30 seconds, or sham therapeutic ultrasound applied to the T4-5 spinal region bilaterally for 30 seconds (the ultrasound machines will not be turned on). Between each of these interventions, subjects will be instructed to rest quietly for five minutes in order to stabilize the body's cardiovagal responses. Following completion of these three interventions, subjects will allowed to ask additional questions and will be given the number of the principal investigator and the IRB office to contact if they have questions or concerns in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* History of back surgeries, osteopenia, osteoporosis, spinal fractures, rib fractures, chronic pain over three months, or heart conditions. Subjects will also be excluded if they are currently taking or have a significant history of taking steroid or anticoagulant medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | 5 minutes pre-intervention (baseline), immediately after each intervention
  Change in heart rate variability monitored continuously

CONTACTS AND LOCATIONS:
Overall Officials: Derrick Sueki, DPT, Principal Investigator — Mount St. Mary's College, Los Angeles, CA
Locations (1):
- Mount St. Mary's College, Los Angeles, California, United States